CLINICAL TRIAL: NCT06768008
Title: Clinical Study of an Integrated Prenatal and Postnatal Treatment Model to Improve the Treatment Effect of Newborns With Critical Congenital Heart Disease
Brief Title: An Integrated Prenatal and Postnatal Treatment Model for the Treatment of Newborns With Critical Congenital Heart Disease
Status: Recruiting | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: Capital Institute of Pediatrics, China (Other); 307 Hospital of PLA (Other)
Responsible Party: Sponsor
Other Study IDs: ZD2024010
Record Dates: First submitted 2024-12-24; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-09

CONDITIONS: Congenital Heart Disease; Coarctation of Aorta; Aortic Stenosis; Pulmonary Atresia; Pulmonary Stenosis; Transposition of the Great Arteries; Truncus Arteriosus; Single Ventricle; Tetralogy of Fallot (TOF); Interrupted Aortic Arch; Hypoplastic Left Heart Syndrome (HLHS); Total Anomalous Pulmonary Venous Connection
Keywords: congenital heart disease; Integrated prenatal and postnatal model; neonate; surgery; Myocardium regeneration
MeSH Terms: conditions — Heart Defects, Congenital; Aortic Coarctation; Aortic Valve Stenosis; Pulmonary Atresia; Pulmonary Valve Stenosis; Transposition of Great Vessels; Truncus Arteriosus, Persistent; Univentricular Heart; Tetralogy of Fallot; Hypoplastic Left Heart Syndrome; Scimitar Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — myocardium, blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

SUMMARY:
The purpose of this two-way cohort study was to explore whether an integrated prenatal and postnatal treatment model for neonates with critical congenital heart disease (CCHD) could be effective in avoiding preoperative morbidities, creating an ideal timing for surgery, thereby reducing postoperative in-hospital mortality, and improving surgical prognosis compared with the traditional model of care. In addition, in neonates with CCHD associated with the right cardiac system, the investigators aim to further investigate whether early postnatal cardiac surgery has the potential advantage of obtaining a time window for myocardial regeneration and thus improving myocardial remodeling. The aim of this study is to improve the diagnostic and therapeutic capacity of critical congenital heart disease and to promote the integrated prenatal-postnatal treatment model for clinical use. This will ultimately improve the quality of healthcare services for patients with cardiovascular diseases and lay the foundation for exploring guidelines for the treatment of cardiovascular diseases suitable for China's national conditions.

The project will be jointly implemented by Beijing Anzhen Hospital , Capital Pediatric Research Institute, and 307 PLA General Hospital. Starting from January 1, 2022, the hospitals will continue to collect hospitalized cases of newborns with CCHD. The integrated prenatal and postnatal model is defined as a definitive diagnosis of CCHD in the fetal period (22-26 weeks), documentation of intrauterine transfer in our obstetrics department, subsequent initiation of an intrapartum or postpartum surgical plan after multidisciplinary consultation, and transfer to the pediatric heart center at the first hour of life, where the child is treated with either postpartum immediate or elective surgery, depending on patient status. For neonates who meet the indications for emergency surgery, surgery is performed immediately after birth. For neonates with non-emergency surgical indications, surgery is performed after birth adjustment to optimal status. The traditional model was defined as postpartum transfer via an outside hospital with routine interventions. The investigators then evaluate surgical prognosis and myocardial regenerative capacity to compare the effects of the two treatment models. This project will validate the advantages of an integrated prenatal and postnatal model over traditional models through real-world research and will improve prognosis in neonates with CCHD.

ELIGIBILITY:
Inclusion Criteria:

1. Full-term infants (gestational age 37-40 weeks): age less than 28 days;
2. Preterm infants (gestational age greater than 32 weeks but less than 37 weeks): corrected gestational age as neonatal period, age less than 28 days;
3. Birth weight > 1.5 kg;
4. Fetal diagnosis of congenital heart diseases by ultrasound at 22-26 weeks of gestation, suitable for biventricular repair.

Exclusion Criteria:

1. Only suitable for palliative surgery or single ventricle repair;
2. Associated genetic/chromosomal abnormalities;
3. Associated with other severe systemic diseases.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with various congenital heart diseases.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of 30-day postoperative mortality | Duration of hospital stay (an expected average of 30 day)
  The purpose of neonatal surgery is to address congenital malformations or other conditions that arise in newborns at birth. Although these surgeries are generally considered safe, there is still a risk of death within 30 days of surgery. Close monitoring and prompt intervention are essential to minimize this risk and ensure the best possible outcome for neonatal patients.

SECONDARY OUTCOMES:
The ratio of neonates received integrated prenatal and postnatal diagnose and treatment | Duration of hospital stay (an expected average of 1 week) and 5 years after discharge]
The incidence of heart failure, metabolic acidosis, severe cyanosis before surgery | Patient status before surgery at hospital
The rate of Medium- and long-term survival rates, and re-operations | During hospitalization (expected to average 1 week) and 5 years post-discharge
  The rate of medium- and long-term survival, as well as the frequency of re-operations, are crucial indicators of the success of surgical interventions. Medium-term survival typically refers to patient outcomes over several months to a few years, while long-term survival indicates the patient's prognosis over many years following surgery. Re-operations may be required due to complications, recurrence of the underlying condition, or failure of the initial surgical procedure. Evaluating these factors helps in assessing the effectiveness of surgical techniques, the quality of patient care, and the need for potential improvements in treatment strategies.

CONTACTS AND LOCATIONS:
Locations (1):
- Biejing Anzhen Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sun Y, Han Y, Li G, Wu Y, Yan J, Wang Q. Prenatal-postnatal integrated management model improves outcomes of neonatal cardiac surgery in critical congenital heart disease: a retrospective cohort study. BMC Pediatr. 2026 Jan 5;26(1):6. doi: 10.1186/s12887-025-06378-x. PMID 41491678